CLINICAL TRIAL: NCT02725112
Title: A Phase 1, Randomized, Open-label, Single-dose, 6-period Study To Investigate The Effect Of In Vitro Dissolution Rate On The In Vivo Bioavailability Of Extended Release Formulations Of Pregabalin In Healthy Volunteers
Brief Title: Bioavailability Study of Pregabalin Extended Release Formulation With Various Release Rates in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A0081309
Record Dates: First submitted 2016-02-10; First posted 2016-03-31 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2017-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Pregabalin ER- Target Release 330mg (Experimental): A: Pregabalin ER tablet formulation, Target release rate, 1 x 330 mg, Oral.
  Interventions: Drug: Pregabalin ER
- Pregabalin ER - Slow Release 330mg (Experimental): B: Pregabalin ER tablet formulation, Slow release rate, 1 x 330 mg, Oral.
  Interventions: Drug: Pregabalin ER
- Pregabalin ER - Fast Release 330mg (Experimental): C: Pregabalin ER tablet formulation, Fast release rate, 1 x 330 mg, Oral.
  Interventions: Drug: Pregabalin ER
- Pregabalin IR - 300mg (Experimental): D: Pregabalin IR capsule formulation, 1 x 300 mg, Oral.
  Interventions: Drug: Pregabalin ER
- Pregabalin ER - Target Release 82.5mg (Experimental): E: Pregabalin ER tablet formulation, Target release rate, 1 x 82.5 mg, Oral.
  Interventions: Drug: Pregabalin ER
- Pregabalin ER - Aberrant Fast 330mg (Experimental): F: Pregabalin ER tablet formulation, Aberrant fast release rate, 1 x 330 mg, Oral.
  Interventions: Drug: Pregabalin ER

INTERVENTIONS:
Drug: Pregabalin ER — A: Pregabalin ER tablet formulation, Target release rate, 1 x 330 mg, Oral.
  Arms: Pregabalin ER- Target Release 330mg
Drug: Pregabalin ER — B: Pregabalin ER tablet formulation, Slow release rate, 1 x 330 mg, Oral.
  Arms: Pregabalin ER - Slow Release 330mg
Drug: Pregabalin ER — C: Pregabalin ER tablet formulation, Fast release rate, 1 x 330 mg, Oral.
  Arms: Pregabalin ER - Fast Release 330mg
Drug: Pregabalin ER — D: Pregabalin IR capsule formulation, 1 x 300 mg, Oral.
  Arms: Pregabalin IR - 300mg
Drug: Pregabalin ER — E: Pregabalin ER tablet formulation, Target release rate, 1 x 82.5 mg, Oral.
  Arms: Pregabalin ER - Target Release 82.5mg
Drug: Pregabalin ER — F: Pregabalin ER tablet formulation, Aberrant fast release rate, 1 x 330 mg, Oral.
  Arms: Pregabalin ER - Aberrant Fast 330mg

SUMMARY:
This study is a Phase 1, randomized, open label, single dose, 6 treatment, 6 period, 6 sequence study in healthy adult volunteers. A total of 24 (4 in each treatment sequence) healthy male and female subjects who, at the time of screening, are between the ages of 18 and 55 years, inclusive will be enrolled. Subjects who discontinue from the study may be replaced at the Sponsor's discretion. Screening activities will be completed within approximately 28 days prior to Day 1 of Period 1. Subjects will be randomized to 1 of the 6 treatment sequences as described in Table 1 below. Each treatment sequence will consist of 6 periods with subjects receiving single doses of pregabalin ER 330 mg target release rate tablet, pregabalin ER 330 mg slow release rate tablet, pregabalin ER 330 mg fast release rate tablet, pregabalin IR 300 mg capsule, pregabalin ER 82.5 mg target release rate tablet, and pregabalin ER 330 mg aberrant fast release rate tablet formulations. All study treatments will be administered following a 600- 750 calorie, 30% fat evening meal.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female subjects and/or male subjects who, at the time of screening, are between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead electrocardiogram (ECG) or clinical laboratory tests. A 1:1 ratio of men to women is desirable, but it will not be considered a protocol deviation if this is not met.
2. Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
3. Evidence of a personally signed and dated informed consent document.
4. Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. History of febrile illness within 5 days prior to the first dose of study investigational product.
3. Subjects with an estimated CLcr <60 mL/min derived using the method of Crockcroft and Gault.1
4. Any condition possibly affecting drug absorption.
5. A positive urine drug screen.
6. Use of tobacco or nicotine containing products in excess of the equivalent of 5 cigarettes per day.
7. History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males (1 drink = 5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) within 6 months of Screening.
8. Treatment with an investigational drug within 30 days or 5 half lives preceding the first dose of study investigational product (whichever is longer).
9. Screening supine blood pressure >= 140 mm Hg (systolic) or >= 90 mm Hg (diastolic), following at least 5 minutes of supine rest. If blood pressure is >= 140 mm Hg (systolic) or >= 90 mm Hg (diastolic), the blood pressure should be repeated 2 more times and the average of the 3 blood pressure values should be used to determine the subject's eligibility.
10. Screening supine 12 lead ECG demonstrating QTc (time from ECG Q wave to the end of the T wave corresponding to electrical systole [QT] corrected for the heart rate) >450 msec or a QRS interval (time from ECG Q wave to the end of the S wave corresponding to ventricle depolarization) >120 msec. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTc or QRS values should be used to determine the subject's eligibility.
11. Pregnant female subjects; breastfeeding female subjects; male subjects with partners currently pregnant; male subjects able to father children and female subjects of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of investigational product.
12. Use of prescription (other than oral, transdermal, intrauterine, implanted, or injected contraceptives or hormone replacement therapy) or nonprescription drugs and dietary supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of study medication.investigational product. Herbal supplements must be discontinued at least 28 days prior to the first dose of study medicationinvestigational product. As an exception, acetaminophen/paracetamol may be used at doses of greater than 1 g/day. Limited use of non prescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case by case basis following approval by the Sponsor.
13. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 56 days prior to dosing.
14. History of sensitivity to pregabalin, gabapentin, or other alpha2 delta ligands.
15. History of sensitivity to heparin or heparin induced thrombocytopenia.
16. Unwilling or unable to comply with the Lifestyle Guidelines described in this protocol.
17. Previous participation in a study involving pregabalin.
18. Subjects who are investigational site staff members directly involved in the study, their family members, site staff members otherwise supervised by the investigator, or subjects who are Pfizer employees directly involved in the study.
19. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2016-02-12 (Actual); Primary Completion 2016-05-22 (Actual); Study Completion 2016-06-17 (Actual)

PRIMARY OUTCOMES:
Cmax from time zero to infinity (AUCinf), when data permits, otherwise AUC from time zero to last quantifiable concentration (AUClast) of pregabalin ER 330 mg slow and fast release rate tablet formulations. | 10 week Study Duration
  To evaluate the relative bioavailability of pregabalin ER 330 mg slow and fast release rate tablet formulations administered immediately following an evening meal.
AUC from time zero to infinity (AUCinf), when data permits, otherwise AUC from time zero to last quantifiable concentration (AUClast) of pregabalin ER 330 mg slow and fast release rate tablet formulations. | 10 week Study Duration
  To evaluate the relative bioavailability of pregabalin ER 330 mg slow and fast release rate tablet formulations administered immediately following an evening meal

SECONDARY OUTCOMES:
Cmax of pregabalin. | 10 week study duration
  To evaluate the PK, safety and tolerability of single doses of pregabalin IR (300 mg) capsule formulation and pregabalin ER (82.5 and 330 mg) tablet formulations in healthy volunteers.
Time to Cmax (Tmax) of pregabalin | 10 week study duration
  To evaluate the PK, safety and tolerability of single doses of pregabalin IR (300 mg) capsule formulation and pregabalin ER (82.5 and 330 mg) tablet formulations in healthy volunteers.
Lag time (Tlag) of pregabalin | 10 week study duration
  To evaluate the PK, safety and tolerability of single doses of pregabalin IR (300 mg) capsule formulation and pregabalin ER (82.5 and 330 mg) tablet formulations in healthy volunteers.
AUC of pregabalin | 10 week study duration
  To evaluate the PK, safety and tolerability of single doses of pregabalin IR (300 mg) capsule formulation and pregabalin ER (82.5 and 330 mg) tablet formulations in healthy volunteers.
Terminal elimination half life (t½) of pregabalin | 10 week study duration
  To evaluate the PK, safety and tolerability of single doses of pregabalin IR (300 mg) capsule formulation and pregabalin ER (82.5 and 330 mg) tablet formulations in healthy volunteers.
Safety endpoints include evaluation of AEs. | 10 week study duration
  To evaluate the PK, safety and tolerability of single doses of pregabalin IR (300 mg) capsule formulation and pregabalin ER (82.5 and 330 mg) tablet formulations in healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New Haven Clinical Research Unit, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081309&StudyName=A%20Phase%201%2C%20Randomized%2C%20Open-label%2C%20Single-dose%2C%205-period%20Study%20To%20Investigate%20The%20Effect%20Of%20In%20Vitro%20Dissolution%20Rate%20On%20The%20In%20Vivo%20Bioavailability%20Of%20Extended%20Release%20Formulations%20Of%20Pregabalin%20In%20Healthy%20Volunteers
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081309&StudyName=A+Phase+1%2C+Randomized%2C+Open-label%2C+Single-dose%2C+6-period+Study+To+Investigate+The+Effect+Of+In+Vitro+Dissolution+Rate+On+The+In+Vivo+Bioavailability+Of+Extended+Release+Formulations+Of+Pregabalin+In+Healthy+Volunteers